CLINICAL TRIAL: NCT01855490
Title: A Pilot Study to Determine the Effects of a Single Dose of Exenatide (Byetta ®) on the Acute Metabolic Responses to a Mixed Meal or Intravenous Glucose Tolerance Test in Patients With Type 1 Diabetes
Brief Title: Study of the Acute Metabolic Effect of Exenatide in Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1201009520
Record Dates: First submitted 2013-01-29; First posted 2013-05-16 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single-arm treatment with Exenatide (Experimental): Exenatide 5 mcg sc. injection 15 minutes prior to a MMTT and IVGTT
  Interventions: Drug: Exenatide

INTERVENTIONS:
Drug: Exenatide

SUMMARY:
The study is designed as an open labeled pilot trial to analyze the acute responses of glucose, GLP-1, GIP, insulin secretory,and glucagon to a mixed meal tolerance test (MMTT) or intravenous glucose tolerance tests (IVGTT) with and without pretreatment with Exenatide (Byetta) 5 mcg sc.

The investigators will also test the effects of Exenatide on gastric emptying during the MMTT.

ELIGIBILITY:
Inclusion Criteria:

* T1D of at least 3 yrs duration.
* Male or female aged 18-56 years who meets the American Diabetes Association standard T1DM criteria.
* HgbA1c<9%
* Insulin requirement of < 0.8 U/kg/d
* Absence of severe hypoglycemia in the past 6 months
* Absence of ketoacidosis in the past 6 months
* Menstruating women must have a negative pregnancy test and be willing to avoid pregnancy during the study period.
* Signed informed consent..

Exclusion Criteria:

* Inability or unwillingness to give informed consent.
* Prior Exenatide or Liraglutide treatment or use of any medication that could potentially affect diabetes or immunologic status
* Known hypersensitivity to Exenatide or any product components
* Participation in an investigational treatment trial within the last 6 weeks before enrollment.
* Any medical condition that in the opinion of the investigator would interfere with safe completion of the trial such as: epilepsy, atopic disease, active Grave's disease, cystic fibrosis, sickle cell anemia, neuropathy, peripheral vascular disease, cerebrovascular disease,liver disease, HIV, or any concurrent autoimmune disease except treated and stable thyroid disease
* Known severe renal impairment, end-stage renal disease or renal transplantation.
* Any history of gastroparesis or other severe gastrointestinal disease, pancreatitis, thyroid nodules or malignancy with the exclusion of a history of localized basal cell carcinoma.
* Uncompensated heart failure, fluid overload, myocardial infarction or liver disease within the last 6 weeks before enrollment.
* Active clinically serious infections.
* Positive pregnancy test in menstruating women or lactating females

Ages: 18 Years to 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2012-01; Primary Completion 2013-07 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Effect of exenatide on metabolic responses to an oral (as a mixed meal) or intravenous glucose challenge in subjects with established T1D with or without residual insulin production. | Each patients is estimated to finish the study within 4-6 weeks
  We will measure the hormonal and metabolic changes during a mixed meal and intravenous glucose tolerance test with and without exenatide pretreatment in subjects with and without residual insulin production.

SECONDARY OUTCOMES:
Effect of exenatide on insulin secretion, glucagon secretion, GLP-1 and GIP levels, and gastric emptying in these patients with T1D. - effect of exenatide on residual insulin production | 4-6 weeks
  In addition to measuring the levels of glucose and gastric emptying, we will measured glucagon levels, insulin secretion rates, GLP-1 and GIP hormonal levels during the provocative tests.

CONTACTS AND LOCATIONS:
Overall Officials: Kevan C Herold, MD, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States